CLINICAL TRIAL: NCT06376370
Title: The Effect of RehaCom Computer-Assisted Rehabilitation Program on Self-Management, Cognitive Function and Quality of Life in Epilepsy Patients: Randomized Controlled Study
Brief Title: The Effect of a Computer-Assisted Rehabilitation Program on Epilepsy Patient
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ülkü Saygılı, Assist. Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16.04.24/2
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy; Computer-assisted Cognitive Rehabilitation; Quality of Life
Keywords: Epilepsy patient; Cognitive rehabilitation; Self management
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): Patients with epilepsy who will receive a computer-assisted cognitive rehabilitation program
  Interventions: Other: Application of computer-assisted cognitive rehabilitation program
- Control (No Intervention): Patients under routine follow-up of the clinic

INTERVENTIONS:
Other: Application of computer-assisted cognitive rehabilitation program — Since the program will respond to the patient's specific needs, the activity may become easier or more difficult depending on the patient's performance. Epilepsy patients will be encouraged by researchers during the exercises and will be able to give feedback on progress at the end of the session. After determining the appropriate time and day for each patient in the experimental group, the intervention will continue for 6 weeks with 45-minute sessions once a week.
  Arms: Study

SUMMARY:
The aim of this study is to examine the effects of the RehaCom Computer-Assisted Rehabilitation Program Applied to Epilepsy Patients on Self-Management, Cognitive Function and Quality of Life.

DETAILED DESCRIPTION:
Modules designed to train cognitive abilities will be used under the supervision of a licensed researcher who is licensed to use the RehaCom application, which is a computer-assisted cognitive rehabilitation program. Researchers can select some modules based on each patient's specific deficits, meaning that deficits can be targeted and specifically trained. Since the program will respond to the patient's specific needs, the activity may become easier or more difficult depending on the patient's performance. Epilepsy patients will be encouraged by researchers during the exercises and will be able to give feedback on progress at the end of the session. After determining the appropriate time and day for each patient in the experimental group, the intervention will continue for 6 weeks with 45-minute sessions once a week.

ELIGIBILITY:
Inclusion Criteria:

* Being registered at Selçuk University Faculty of Medicine Hospital Neurology Polyclinic
* Having been diagnosed with epilepsy for at least 6 months
* Being between the ages of 18 and 60 (60 is the age limit for the Moxo test)
* Volunteer to provide transportation to Selçuk University Faculty of Medicine for research one day a week.
* Ability to use tools such as computer mouse and telephone
* Score 24 or more from the Mini Mental State Test

Exclusion Criteria:

* Individuals have physical, mental, visual and hearing disabilities
* Having another neurological disorder
* The individual has a transportation disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Test | 5 minutes
  Mini-mental state test (MMSE), a simple screening test, is a useful test that indicates cognitive impairment and is also used in follow-up.The mini mental state assessment test developed by Folstein et al. (1975) is a test that measures patients' orientation, memory, attention and calculation, recall, language, motor function and perception aspects and is evaluated out of 30 points. It is accepted that cognitive status worsens as the scores patients receive decrease. Although the test has limited specificity in terms of distinguishing clinical syndromes, it is a short, useful and standardized method that can be used to determine the cognitive level globally.
Epilepsy Quality of Life Scale | 10 minutes
  The validity and reliability study of the E-31 Scale and the QOLIE-89 Scale in our country was conducted by Mollaoğlu et al. It is a scale consisting of 31 items out of 89 items in the QOLIE-89 Scale made by. In the QOLIE-31 Scale, only epilepsy-related issues are questioned. QOLIE -31 scale consists of 7 sub-dimensions including the following health concepts. These sub-dimensions; seizure-related concerns (5 items), emotional well-being (5 items), energy/fatigue (4 items), social function (5 items), cognitive function (6 items), effects of medications (3 items), total quality of life (2 items). It consists of a total of 31 items, including an additional item assessing total health status. The QOLIE-31 Scale, which normally consists of 30 items, has gained the feature of a 31-item scale with the addition of this last item (the item that evaluates the total health status). The scale is scored between 0-100. A high score reflects a high quality of life.
MOXO Test | 18 minutes
  MOXO Adult is a computerized, distractor-continuous performance test, an objective tool that measures a person's attention profile. The MOXO Adult test includes distractor systems that establish a connection with the person's environment. MOXO continuous performance test is a measurement tool designed to diagnose symptoms related to attention and cognitive status, with scientifically proven sensitivity (90%) and specificity (85%). The test is an 18.2-minute test consisting of eight blocks (53 trials in each block). On each trial, a stimulus (target or nontarget) is presented in the center of the computer screen. This is followed by a "gap" of the same period in which no stimulus is presented. Participants are asked to press the space bar in response to targets and to refrain from pressing it in response to nontargets. This is done by ignoring a number of visual and auditory distractions.
Epilepsy Self-Management Scale | 12 minutes
  The Epilepsy Self-Management Scale was developed by Dilorio et al. (2004) mainly to evaluate the frequency of use of epilepsy self-management practices or behaviors. The validity and reliability study of the scale was conducted by Yeni et al. (2020). This scale, consisting of 38 items, has five subsections that evaluate medication (10 items), information (8 items), safety (8 items), seizure (6 items) and lifestyle (6 items) management in epilepsy patients. Responses are evaluated in a 5-point Likert format and scored between 1-5. Scoring is done on a frequency scale, where 1 is "never" and 5 is "always". There are also reverse coded items in the scale, and these are converted to their normal form during the evaluation and included in the process. The minimum score that can be obtained from the scale is 38 and the maximum score is 190, and high scores indicate that patients have good self-management.

CONTACTS AND LOCATIONS:
Locations (1):
- ülkü Saygili Düzova, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No